CLINICAL TRIAL: NCT01142960
Title: Effects of Lycium Barbarum Supplements on the Progression of Senile Cataract in Hong Kong Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Chea-su Kee, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5-ZH73
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Lens Opacity
MeSH Terms: conditions — Cataract | interventions — Starch; lycium barbarum polysaccharide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Active Comparator): Starch
  Interventions: Dietary Supplement: Starch
- Lycium Barbarum (Experimental): Lycium Barbarum supplement
  Interventions: Dietary Supplement: Lycium Barbarum

INTERVENTIONS:
Dietary Supplement: Starch — 1350mg/day
  Arms: Placebo
Dietary Supplement: Lycium Barbarum — 1350mg/day
  Arms: Lycium Barbarum

SUMMARY:
With the rapid growing aging population, age-related eye diseases including cataract are becoming more prevalent. The demand for cataract surgery and post-surgical care posed enormous financial burdens to the government.

Lycium barbarum contains lutein and zeaxanthin which can filter the phototoxic blue light and neutralize the reactive oxygen species, thus provide a protective effect against cataract formation.

This study aims to determine the effects of Lycium barbarum Supplements on the progression of senile cataract in Hong Kong Chinese elderly.

DETAILED DESCRIPTION:
Please note that a manuscript for this study is being prepared. Detailed description will be provided after we come up with the final draft.

ELIGIBILITY:
Inclusion Criteria:

* Unlikely to have cataract surgery within 3 years
* Presence of mild to moderate cataract in one or both eyes, graded by Lens Opacities Classification System III (LOCSIII).
* logMAR acuity equivalent to Snellen acuity of 20/63 or better
* no previous history and clinical signs of glaucoma by determining intraocular pressure using applanation Tonometry (no more than 22mmHg)
* no ocular anomalies: amblyopia, binocular anomalies, ocular trauma
* no history of eye surgery, laser treatment, iritis, retinal crystalline deposits, macular degeneration, or optic nerve diseases
* no extended use of systemic or ocular corticosteroid drugs
* no concurrent participation of other systemic or ocular drug intervention study

Exclusion Criteria:

* diabetes mellitus
* renal failure
* fat malabsorption syndrome
* intestinal surgery history
* chronic diarrhea
* alcoholism
* use of anticoagulants
* regular use of nutritional supplements such as multi-vitamin, mineral and other antioxidant supplements (including Omega-3)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Lens Opacity Classification System III (LOCSIII) | 3 years

SECONDARY OUTCOMES:
Visual Acuity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chi-wai Do, PhD, Principal Investigator — The Hong Kong Polytechnic University; Chea-su Kee, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided